CLINICAL TRIAL: NCT02946567
Title: Game to Improve Hearing Health Care Outcomes
Acronym: NoisyCity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Photozig, Inc. (Industry)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Bruno Kajiyama, CEO, Photozig, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pz-A105a; R44DC013114 (NIH)
Record Dates: First submitted 2016-10-24; First posted 2016-10-27 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Focus of the Study is to Promote Healthy Hearing

ARMS (2):
- Noisy City (Experimental): Participant will play the Noisy City game developed by this project.
  Interventions: Other: Noisy City information about hearing health care
- Control (Placebo Comparator): Participant will play a generic game.
  Interventions: Other: Generic Game

INTERVENTIONS:
Other: Noisy City information about hearing health care — Participants will play the game Noisy City, which contains information about hearing health care.
  Arms: Noisy City
Other: Generic Game — Participants will play a generic game without any particular information about hearing health care.
  Arms: Control

SUMMARY:
The investigators are studying the educational potential of games, with the goal of developing a game to improve learning and promote healthy hearing behaviors.

The project is looking for adolescents and young adults that play games to share their experience and learning from playing games.

The investigators ask participants to fill out an enrollment form/informed consent, complete surveys on healthy hearing habits, and play a game provided by the project.

This projects aims the development and evaluation of a game to educate teenagers and young adults about noise-induced hearing loss, enhance knowledge about hearing, and promote healthy hearing behaviors with the potential to improve hearing health care.

ELIGIBILITY:
Inclusion Criteria:

* Participants have to be between the ages of 13 and 20 years of age (either gender).
* Participants who are between the ages of 13 and 17 years of age must have a willing and able parent or legal guardian who permits them to participate.
* Participants must have Internet access, an email address (or be able to use parent's/legal guardian's email address), and agree to play a game (random assignment to a group with a different game).

Exclusion Criteria:

* Participants will be excluded if they are cognitively impaired, have any serious medical problem that may interfere with their ability to engage with the online game.
* Those who are not able to read/follow written instructions and individuals with an excessive addiction to games will be excluded.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Knowledge, Attitudes, and Intended Behavior Questionnaire about hearing health care | 9 weeks
  This instrument has been used to evaluate the effectiveness of past hearing loss prevention programs funded by the National Institute of Health. It contains questions on knowledge, attitudes, and intended behavior related to hearing health care. Although there are questions in different domains, the instrument consolidates the overall perception of participant on hearing health care.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Kajiyama, MS, Principal Investigator — Photozig, Inc.
Locations (1):
- Photozig, Inc., Moffett Field, California, United States